CLINICAL TRIAL: NCT03436875
Title: Cardiometabolic Health in Adult Latinos in the Rio Grande Valley With and Without Specific Gene Mutations
Brief Title: Cardiometabolic and Mental Health in the RGV
Status: Withdrawn | Type: Observational
Why Stopped: Pause for preliminary data analysis
Sponsor: University of Texas Rio Grande Valley (Other)
Responsible Party: Principal Investigator, Ryan Russell, Assistant Professor, University of Texas Rio Grande Valley
Other Study IDs: 2017-094-04
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Microvessels; Carbohydrate Metabolism; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected during an oral glucose tolerance test. Plasma will be stored in -80 for later testing (insulin, cytokines, etc). Buffy coat will also be stored at -80 for specific SNP analysis for likely candidate genes affecting microvascular blood flow and impaired substrate oxidation. Stool samples will be collected to asses the microbiota.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: Healthy people either with (FH+) or without (FH-) a family history of diabetes or Alzheimer's Disease.
- unhealthy: People type 2 diabetes or Alzheimer's Disease that have either: a family history of that disease (FH+) or no family history of T2D or Alzheimer's for two generations (FH-).

SUMMARY:
Microvascular insulin resistance has been shown to precede myocyte insulin resistance and impairments in metabolic function. However, there is no convincing data showing the relationship between impaired microvascular flow and impaired metabolic flexibility. Recent evidence exists that impaired microvascular blood flow in Caucasians directly contributes to impaired metabolic flexibility in Caucasians (Diabetes Care), however there is no such evidence in Hispanics. Since there is a large disparity in cardiometabolic disease in Hispanics, this study aims to determine the role of impaired microvascular blood flow on impaired substrate oxidation switching (metabolic flexibility) in healthy people at risk for developing type 2 diabetes.

DETAILED DESCRIPTION:
Metabolic flexibility is the ability to adjust fuel oxidation to fuel availability. The term is classically defined as the ability to switch from fat oxidation during fasting conditions to glucose oxidation during insulin stimulation (e.g. a meal, OGTT, or hyperinsulinaemic euglycaemic clamp). It is well established that people with insulin resistance and T2D are not metabolically flexible, thus do not switch oxidized fuels as efficiently as insulin sensitive individuals. However, simply looking at fasting respiratory exchange ratio (RER) is not adequate, as fasting fat oxidation can sometimes increase with the progression of T2D , lowering RER. Furthermore, people with the same fasting RER can have different degrees of metabolic flexibility, as we previously shown (Figure 5). Factors thought to mediate MF have been eloquently outlined in a perspective piece. In general, impaired MF is proposed to be caused by over-nutrition, leading to over-supply of main substrates (glucose, lipid, and amino acids) to the mitochondria, leading to disruption of signaling events mediating glucose/fatty acid oxidation switching originally proposed by Randle and colleagues. Of particular interest to this perspective of impaired MF is the requirement of either insulin resistance, or the necessity of being in a state of positive energy balance. As Dr. Russell has previously shown (Figure 5), FH+ people display similar fasting RER/RQ, but impaired MF similar to those with T2D, but with no signs of insulin resistance nor over-nutrition (as these participants were healthy, lean collegiate athletes and their collegiate athletic trainers). These data suggest that healthy FH+ develop/display impaired MF though completely different means than the current body of literature can explain. In addition, as noted in Figure 4, re-testing a similar cohort (healthy FH+/-) to compare OGTT vs MMC indicates that glucose excursions present in FH+ during the MMC are masked during an OGTT, suggesting that the MMC is more sensitive than an OGTT at detecting variations in glycemic and MBF regulation.

Skeletal Muscle Microvascular Blood Flow helps to regulate glucose disposal by increasing delivery of glucose and insulin to the myocytes. Loss of normal microvascular function is an early driver in the development of muscle insulin resistance, indicating an early therapeutic target for prevention of insulin resistance within muscle. Blocking this microvascular action of insulin (e.g. with vasoconstrictors, inflammatory cytokines, or elevated FFAs) directly cause muscle and whole body insulin resistance [8]. This microvascular action of insulin is lost during pre-diabetes and T2D in humans, though can be improved with resistance training. As there is a strong connection between skeletal muscle microvascular responses, and metabolic function (glycemic regulation and metabolic flexibility - Figure 1), we anticipate that healthy FH+ will also display impaired MBF in response to a MMC, partially explaining their metabolic dysfunction. The importance of using contrast-enhanced ultrasonography (CEU) to detect changes in MBF in real time is extremely valuable, and is discussed in the recent editorial by Dr. Linder about our April 2018 CEU paper MBF changes in adipose tissue.

Macrovascular Responses. Large blood vessel function is correlative to risk of developing hypertension and cardiovascular disease. Large blood vessel function can be measured in a number of ways including insulin-mediated dilation (degree of brachial artery dilation following an OGTT) using 2D and Doppler ultrasound. Dr. Russell has expertise in this technique in healthy, obese, and T2D populations and found that responses are improved with RT.

Recent studies from the Framingham Heart Study have indicated that large artery (aortic) stiffness precedes hypertension. Measurement of carotid-to-femoral pulse wave velocity (by applanation tonometry) is the gold standard technique to assess central artery stiffness. Drs. Russell and Karabulut have expertise in these techniques demonstrating pathologies associated with arterial stiffness.

Oral Glucose Tolerance Test (OGTT). Overnight fasted participants will undergo an OGTT in order to determine glucose tolerance intolerance. A catheter will be placed into a median deep antecubital vein for blood sampling. Each participant will consume 75g of glucose. Plasma glucose will be measured while fasting, and at 15, 30, 60, 90, and 120 min following the glucose load to measure the time course for glucose appearance/disappearance. Plasma proinsulin, insulin, C-peptide and glucagon will be measured at these times to assess pancreatic function. We will also measure glucagon-like peptide-1 (GLP-1).

Mixed Meal Challenge (MMC). A catheter will be placed into a median deep antecubital vein on one arm for blood sampling. Each subject will receive a liquid mixed meal (299 calories - 42 from fat, 144 from carbohydrate, and 113 from protein). Blood sampling and analysis with MMC will be as described above for the OGTT.

METABOLIC & VASCULAR MEASURES (Conducted during OGTT/MMC). Whole body RER and Metabolic Flexibility. Metabolic flexibility will be determined via indirect calorimetry by quantifying changes in oxidation of lipid and carbohydrate (via RER changes) from fasting through 60-minutes after consumption of the OGTT and MMC. Briefly, a canopy will be placed over the heads of the participants which will be attached to an indirect calorimetry metabolic cart equipped for resting metabolic rate (RMR) measures (ParvoMedics TrueOne 2400) to analyse breath gas in a semi-recumbent position. After a 20-minute acclimatization period, breath gas data will be collected continuously for 30 min prior to the OGTT and MMC. Following RMR, the OGTT or MMC beverage will be consumed by the participant (within 2 minutes), and then the canopy will be replaced over their head for 60-min post OGTT/MMC consumption. Changes between fasting, and during OGTT/MMC testing will be used to calculate substrate oxidation and metabolic flexibility as done previously by the PI.

Skeletal Muscle Microvascular Perfusion. Dr. Russell was trained for two years in the field of contrast enhanced ultrasonography (CEU) by Dr. Keske, a world leader in CEU imaging of skeletal muscle. CEU imaging of forearm muscle will be performed using an L9-3 linear array transducer interfaced to an iU22 ultrasound (Philips) during microbubble (Lumison®) infusion as described previously [17, 18]. CEU images will be analysed off-line using Qlab (Version 10.8, Philips) to determine microvascular blood volume (A), microvascular flow velocity (β) and microvascular perfusion (A×β) as done previously by the PI. These MBF responses in muscle will be assessed at rest and 1hr into the OGTT and MMC as done previously (Figure 1).

Macrovascular Responses. Brachial artery diameter and blood flow velocity will be determined proximal to the antecubital fold using a high frequency L12-5 linear array transducer interfaced to an iU22 ultrasound (Philips Medical Systems). Brachial artery responses will be measured at baseline and 1-hr following the OGTT/MMC which will determine insulin sensitivity of large blood vessels.

Central and Peripheral Hemodynamics. Brachial blood pressure will be measured using automated blood pressure devices while fasting, and again 60-min post OGTT/MMC. Central blood pressure and arterial stiffness will be determined using SphygmoCor tonometry as done previously. Briefly, the subjects will lie down in the supine position for a minimum of 10 minutes, and baseline arterial elasticity and hemodynamics will be measured using hypertension diagnostic (noninvasive equipment conducts measurements of arterial stiffness via placing a sensor on the radial artery at the right wrist and a cuff to the left arm to measure blood pressure) and measurement of pulse wave velocity using SphygmoCor (which is conducted noninvasively using a pulse wave velocity analyzer in segmental measures at the carotid, femoral, and the dorsalis pedis while wearing three electrodes on the chest to monitor the heart's electrical activity).

Large artery stiffness. Aortic pulse wave velocity (PWV) will be recorded by sequential applantation tonometry (SphygmCor) at carotid and femoral arteries as described previously. Large artery stiffness will be measured at baseline and 1-hr following the OGTT/MMC and will inform us of how stiff these large blood vessels are, which can predict risk of hypertension and CVD.

Specific Aim 2. In order to identify novel physiological mechanisms whereby RT program improve indices of metabolic function and muscle microvascular responses, OGTT and MMC testing from Aim 1 will be repeated after a 6-week RT intervention in all participants - T2D and healthy, FH+ and FH-. As discussed above, having a family history of T2D increases risk for developing T2D than FH-, which may result from early impairments in MF [5]. The pathology behind impaired MF is not fully understood, though is thought to occur early in the cardiometabolic continuum as it occurs concomitant with impaired MBF responses in skeletal muscle, both of which manifest prior to glucose intolerance. Although exercise training has been shown to improve lipid oxidation relevant to impaired MF, the effect of exercise on MF is unclear. In a classical study using interventions to 1) increase physical activity, and 2) decrease physical activity with bed rest, in combination with cross-sectional analysis of fit and unfit humans indicate a strong positive relationship between physical activity and MF. Further, there is convincing translational data to indicate that higher MF noted in trained vs. untrained humans (cross-sectional) may be due to the mobilization and reesterification of intramyocellular triacylglycerol (IMTG) and improved lipid partitioning. However, neither of these studies accounted for a family history of T2D. Yet, preliminary data for this application indicate that healthy FH+ are metabolically inflexible, in spite of regular participation in exercise. This phenomenon further supports the notion that the etiology of impaired MF in FH+ deviate from traditional mechanisms affecting MF.

The beneficial effects of exercise training on vascular health have been extensively reviewed. Further, we have shown that RT lowers fasting blood glucose in healthy FH+ and FH- alike, and that RT improves glycemic regulation concomitant with improve skeletal muscle MBF. The improved glycemic and microvascular regulation we noted are supported by recent work indicating that increased insulin sensitivity and glucose disposal noted post-exercise are the result of increased insulin-stimulated phosphorylation of Akt and enhanced activation of glycogen synthase, but only in combination with concomitant increase skeletal muscle MBF. Additionally, a recent publication in Circulation indicates exercise may override genetic factors associated with increased risk of cardiovascular disease. Therefore, an important step beyond Aim 1 is to elucidate physiological mechanisms whereby RT improves cardiometabolic health, specifically in FH+ Hispanics.

The effects of exercise training in the FH+ population is of particular interest, as beneficial health benefits of exercise interventions in FH+ are not uniform. As noted in Figure 2, preliminary data from the PI suggests that FH+ people with T2D may have greater improvements in glycemic regulation and MBF responses than their FH- counterparts. This is in contrast to work done by Ekman showing that FH- had greater improvements in expression of genes involved with metabolism, oxidative phosphorylation, and cellular respiration than FH+. Notably, these differences were noted only while controlling for total exercise performed (quantified by energy expenditure during exercise), of which, FH+ performed 61% more than FH-. Taking on a different perspective, these findings suggest that FH+ actually have greater improvements in cardiometabolic function with training because they perform more exercise ad libitum than matched FH-. Taken together, we hypothesize that RT will markedly improve our microvascular and metabolic measures more in FH+ than FH-, independent of T2D status.

Innovation. Combining gold-standard microvascular techniques with metabolomics and measures of metabolic flexibility in order to identify novel mechanisms of cardiometabolic function that relate to disease onset and progression, and also to reversal with exercise training fills a much-needed gap in our understanding of cardiometabolic disease. Performing this study in Hispanics of the RGV with and without a family history of T2D is a novel and feasible integration of: 1) early detection of cardiometabolic disease, 2) physiological mechanisms of improved cardiometabolic function with exercise, and 3) health disparities research. We know exercise improves cardiometabolic health. However, by including an exercise intervention with our novel testing approach, we not only identify early pathophysiological markers of cardiometabolic disease, but we can also learn the degree to which these physiological processes improve. This is vitally important in identifying potential mechanisms for targeted therapy. For example, if MBF responses and glycemic regulation improve, but not MF, it is possible that impaired MF in the FH+ population may not be a metabolic defect, and thus not a viable target for treatment. This approach to identify specific early physiological mechanisms of cardiometabolic disease that change with exercise training can refine therapeutic targets, potentially alleviating a huge financial burden on the healthcare system, and reducing cardiometabolic disease disparities.

Resistance Exercise Program. This 6-week RT program will be conducted as done previously by the PI. Briefly, RT will be done 3 days/week, and consist of: 1) a pre-training week (three 1-hour sessions) for participants to learn exercise movements, gym safety, and proper lifting form, and to calculate of the weight each participant can lift in a single repetition (1-RM) ; 2) a 6-week RT program including plyometrics and core. The RT program will include weight training 2 days per week (with at least 2 days of rest between) and plyometrics/core done 1 day per week (not on a weight training day) with all exercise supervised by Dr. Russell. Exercise will be the same between FH+ and FH- groups. Weight lifting exercises include: squat (or leg press, depending on ability), bench-press, lateral pull-down, seated row, shoulder press, push-up, bicep curl, triceps extension, dead-lift, and abdominal exercises. Training progression will be continuously monitored and load adjusted to ensure that each participant increases the resistance load with increasing strength, enabling them to work at 65-85% of 1-RM for each workout. Plyometrics will start as low-impact, and progressively become more challenging as fitness improves. These include: squat jumps, lunge jumps, box jumps, various medicine ball techniques, and shuttle runs. Exercise sessions will take approximately 40-50 min, including a warm-up/cool-down period. The PI has shown that this type of RT program is effective at lowering fasting blood glucose in healthy FH+, and improving MBF responses and glycemic control in those with T2D [23].

This study utilizes a pre/post intervention randomized cross-over study design in that OGTT and MMC testing will be administered in random order both before, and after RT. Since acute exercise is known to influence outcomes pertinent to this application, post-RT testing in the first randomized test (either OGTT or MMC) will be performed between 48 and 56 hours after the last RT session. Further, the second post-RT test (either OGTT or MMC not used in the 1st test) will be scheduled 1 week later. To ensure detraining does not affect outcomes, two more interim training sessions will be conducted in the week between post-RT tests 1 and 2, with the second post-RT test day occurring between 48 - 56 hours after the last interim RT session.

Specific Aim 3. In order to determine associations of microvascular and metabolic function with metabolomic profiling in Hispanics with and without a family history of T2D, we are testing people with and without T2D, in a population with stratified cardiometabolic disease risk (FH+ and FH-). Metabolomic profiling via gas Chromatograph Time-of-Flight Mass Spectrometer (GC×GC-ToFMS) will be performed to identify various lipid and amino acid sub-species (acyl-carnitines) in serum: 1) before RT (fasting, and 60-min after OGTT/MMC), and 2) after RT (while fasting, and 60-min after OGTT/MMC).

ELIGIBILITY:
Inclusion Criteria:

* Healthy people, those with T2D, or those with Alzheimer's Disease.
* 18-75 years
* having either a parent with type 2 diabetes or Alzheimer's, or no history for 2 generations
* non-smoking, weight-stable

Exclusion Criteria:

* presence of microvascular disease
* smoking
* having gained or lost more than 5lbs in the last 3 months
* pregnancy
* having cancer, liver, or kidney disease within 5 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Hispanics residing in Southeast Texas ages 18 - 70 years old that have either a parent with type 2 diabetes or Alzheimer's, or no history of type 2 diabetes or Alzeimer's for two generations.
  People with type 2 diabetes or Alzheimer's and controlled hypertension that have either: a parent with type 2 diabetes, or no history of type 2 diabetes for two generations.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Microvascular responses in skeletal muscle | 4 years
  Changes in microvascular blood flow in skeletal muscle from fasting to post-OGTT or post-MMC.
Microbiota | 4 years
  Classification of microbiota to determine its impact on cardiometabolic and mental health

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Rio Grande Valley - Cardiometabolic Exercise Lab, Brownsville, Texas, United States

IPD SHARING:
Plan to Share IPD: No